CLINICAL TRIAL: NCT03586141
Title: Validation of Hb-measurement of Pronto ® as Screening Tool for Preoperative Diagnostic of Anemia
Brief Title: Pronto for Patient Blood Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Dr. Eva Wittenmeier, Principal Investigator, Johannes Gutenberg University Mainz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pronto for PBM
Record Dates: First submitted 2018-06-21; First posted 2018-07-13 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: measurement of hemoglobin by a noninvasive sensor clip
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- noninvasive measurement of hemoglobin (Other): All participating patients are measured by the Pronto® hemoglobin measurement tool
  Interventions: Diagnostic Test: Pronto® hemoglobin measurement tool

INTERVENTIONS:
Diagnostic Test: Pronto® hemoglobin measurement tool — All patients who are planned to undergo elective surgery come to the preoperative anesthetic ambulance. They are all measured by the Pronto® hemoglobin measurement tool

SUMMARY:
The concept of Patient Blood Management requires preoperative diagnostic of anemia. To avoid the harmful procedure of venous puncture for drawing a blood sample, noninvasive measurement of hemoglobin has been developed. However noninvasive measurement of hemoglobin has yet been not accurate enough to replace invasive hemoglobin measurement. This study investigates if a noninvasive measurement tool can serve as a screening tool to find out for which patients invasive measurement of hemoglobin is necessary.

DETAILED DESCRIPTION:
The noninvasive hemoglobin measurement tool Pronto® can measure hemoglobin noninvasively by a sensor clip. The investigators analyzed previous studies with the Pronto device and calculated two cut-off values of the noninvasive hemoglobin device. If noninvasive hemoglobin values are higher than cut off value 1 the investigators postulate that with a sensitivity of 99% the participant has no anemia. To confirm this, participants who are supposed to undergo elective surgery and come to the preoperative anesthetic ambulance are measured by the Pronto-device. The noninvasive measurements are compared with the laboratory values of the patients and cut-off value 1 can be confirmed.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children >=3kg that are planned to undergo elective surgery
* Written informed consent

Exclusion Criteria:

* no written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1129 (Actual)
Dates: Start 2018-07-22 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Validation of a postulated noninvasively measured haemoglobin value as a cut-off value for the decision wether invasively measuring of haemoglobin concentration for preoperative patient blood management is necessary. | five to ten minutes
  Previous studies show that noninvasively measured haemoglobin is not accurate enough to determine exactly the haemoglobin value for preoperative diagnosis of anaemia. We postulate that noninvasive haemoglobin measurement can be used as a screening tool to decide wether invasive measurement of haemoglobin is necessary. We calculated a cut-off value 1 by analysing previous studies. Noninvasive haemoglobin measurements that are above the cut-off-value are postulated to show that the patient is not anaemic with a sensitivity of 99%.

SECONDARY OUTCOMES:
Validation of postulated non invasively measured haemoglobin value as a cut off-value 2 | five to ten minutes
  We calculated a cut-off value 2 by analysing previous studies. Noninvasive haemoglobin measurements that are below the cut-off-value 2 are postulated to show that the patient is anaemic with a speciality of 99%.
Agreement between invasive and noninvasive measurement in adults and children | five to ten minutes
  Noninvasive haemoglobin measurement values are compared with invasive haemoglobin measurement values

CONTACTS AND LOCATIONS:
Overall Officials: Eva Wittenmeier, MD, Principal Investigator — Johannes Gutenberg University Centre, department of anaesthesiology, Langenbeckstraße 1, 55131 Mainz, Germany
Locations (1):
- Johannes Gutenbert University Centre, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohnke K, Smetiprach J, Paumen Y, Mildenberger P, Komorek Y, Griemert EV, Wittenmeier E. Is noninvasive hemoglobin measurement suitable for children undergoing preoperative anesthesia consultation? J Clin Monit Comput. 2025 Feb;39(1):175-182. doi: 10.1007/s10877-024-01194-7. Epub 2024 Jul 20. PMID 39031232
- [Derived] Wittenmeier E, Paumen Y, Mildenberger P, Smetiprach J, Pirlich N, Griemert EV, Kriege M, Engelhard K. Non-invasive haemoglobin measurement as an index test to detect pre-operative anaemia in elective surgery patients - a prospective study. Anaesthesia. 2021 May;76(5):647-654. doi: 10.1111/anae.15312. Epub 2020 Nov 23. PMID 33227153